CLINICAL TRIAL: NCT00144976
Title: Pilot Study, Without Direct Individual Benefice, of Biological Effect of Tarceva (OSI-774) at Posology of 150 mg by Day for Patients Stricken by ENT Epidermoid Carcinoma Waiting for First Surgical Picking up.
Brief Title: Study of Biological Effect of Tarceva (OSI-774) for Patients Stricken by ENT Epidermoid Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Dr Jean-Pierre DELORD, Institut Claudius Regaud
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 03 VADS 01
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2008-05

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms; Tarceva; ENT
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tarceva — Tarceva will be administered at dosage 150 mg od one hour before or two hours after meat. Patients will receive Tarceva between 18 and 28 days.
  Other Names: erlotinib

SUMMARY:
The purpose of this study is to evaluate the biological effect of Tarceva (OSI-774) from an inhibition of EGF tumor receptor tyrosine kinase activity's point of view, for patients who are carriers of head and neck epidermoid carcinoma.

DETAILED DESCRIPTION:
Patients will receive Tarceva in continuous between 18 and 28 days after pan-endoscopy exam until surgery

ELIGIBILITY:
Inclusion Criteria:

* Neck and head epidermoid carcinoma histologically proved. Patient with an ENT epidermoid tumor can be included in the study if this relapse is located in an area not irradiated yet.
* At least tumor classified T2NXM0
* Patient who can be picked up in a first surgery with a curative purpose or who must have a necessity's surgery (cervical curettage for voluminous adenopathies before radiotherapy)
* Patient without clinical or radiological sign of metastatic disease
* Good general status (OMS ≤ 2)
* Patient able to ingest food.
* Age ≥ 18 years
* Well-informed written consent, signed by the patient.
* Patient with sickness benefit

Exclusion Criteria:

* Patient with relapse ever treated by radiotherapy
* Other prospective study's participation
* Recent and massive digestive haemorrhage
* Medical contra-indication like main general status alteration, uncontrolled serious infectious disease, main uncontrolled metabolic anomaly ongoing.
* Pre-existent pulmonary pathology (BPCO, pleurisy, lymphangitis, interstitial syndrome)
* Severe cardiac pathology (stage 3 or 4 cardiac insufficiency, unstable angina pectoris, uncontrolled arrhythmia, myocardium's infarction antecedent during the year that precede the inclusion.
* Ophthalmic pathology antecedent concerning the ocular surface or lens-carrier
* Concomitant administration, by local or general tract, of drug responsible for ocular drought or which could delay the epithelial cicatrization
* Less than 1000 polynuclear neutrophil leucocytes or less than 75000 blood-platelets at inclusion
* Bilirubin at higher concentration than one point five times the normal
* Renal insufficiency (glomerular filtration flow ≤ 40 ml/min)calculated in accordance with Cockroft's formula
* Tacking of Beta blockers, amiodarone, NSAIDs, bleomycin, just before or during the study
* Pregnant or nursing women
* Patient under guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the biological effect of Tarceva (OSI-774) from an inhibition of EGF tumor receptor tyrosine kinase activity's point of view, for patients who are carriers of head and neck epidermoid carcinoma.

SECONDARY OUTCOMES:
Correlation study between pharmacokinetic and biological effect observed of molecule OSI-774.
Verification of biological effect of Tarceva's homogeneity (inhibition of EGFR-TK) according to sites, particularly from the point of view of a possible difference primary tumor/metastatic adenopathy and tumorous tissue/healthy tissue.
Characterisation of OSI-774 modes of action from the cellular cycle arrest proteinic effectors's point of view.
Constitution of frozen tissue bank for genomic (sequencing) study of tumorous EGF-R structure and for modification of in situ gene expression induction with OSI-774 by RNA microarrays technology.
Pharmacogenomics study of Tarceva's metabolism : genes studied code for cytochrome 3A5 and glycoprotein-P.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Delord, Docteur, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - Center Oscar Lambret, Lille
  - Institut claudius regaud, Toulouse